CLINICAL TRIAL: NCT01372800
Title: Serum Adiponectin Concentration, Activity and Isoforms in Chinese Population and Its Correlation to Cardiovascular and Cerebrovascular Diseases
Brief Title: Serum Adiponectin in Chinese Population and Its Correlation to Cardiovascular and Cerebrovascular Diseases
Status: Recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: xj050503
Record Dates: First submitted 2011-06-10; First posted 2011-06-14 (Estimated); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Myocardial Infarction; Cerebral Infarction
Keywords: adiponectin; cardiovascular diseases; cerebrovascular diseases
MeSH Terms: conditions — Myocardial Infarction; Cerebral Infarction; Cardiovascular Diseases; Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- volunteer

SUMMARY:
Adiponectin (Ad) is an abundant protein in human body, and reports have shown that it act as a novel risk factor for brain and heart ischemia injury. This 5 years follow-up study will focus on serum adiponectin concentration, activity and isoforms in Chinese population and its correlation to these diseases.

DETAILED DESCRIPTION:
Adiponectin (Ad) is an abundant protein hormone regulatory of numerous metabolic processes, anti-inflammatory, vascular protective, and anti-ischemic properties. Since its 1995 discovery, Ad has garnered considerable attention for its role in diabetic and cardiovascular pathology. Clinical observations have demonstrated the association of hypoadiponectinemia in patients with obesity, cardiovascular disease, and insulin resistance. There is growing evidence supporting Ad can act as a novel risk factor for cardiovascular and cerebrovascular injury. This 5 years follow-up study will focus on serum adiponectin concentration, activity and isoforms in Chinese population and its correlation to cardiovascular and cerebrovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

* available for 5 years of follow-up study

Exclusion Criteria:

* Death caused other than cardiovascular and cerebralvascular diseases till the study ends
* Floating Population
* Pregnancy, lactation, or child bearing women
* Tumor
* Active hepatic disease or hepatic dysfunction, or AST/ALT > 1.5UNL
* Severe renal dysfunction(Scr > 3 mg/dl or 264μmol/L)
* Patients with any condition which, in the investigator's judgment, might increase the risk to the subject for any adverse event or abnormal laboratory finding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: volunteer
Sampling Method: Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2011-05-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2036-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with major adverse events | 5 years
  Major adverse events included but were not limited to death during the study caused by cardiovascular events or cerebrovascular events.

SECONDARY OUTCOMES:
blood routine, glucose and lipid profile; ECG; | 5 years
  the tests mentioned above will be taken once per year
serum adiponectin concentration, activity and isoforms | 5 years
  serum adiponectin concentration, activity and isoforms will be monitored once per year.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Gao C, Zhao S, Lian K, Mi B, Si R, Tan Z, Fu F, Wang S, Wang R, Ma X, Tao L. C1q/TNF-related protein 3 (CTRP3) and 9 (CTRP9) concentrations are decreased in patients with heart failure and are associated with increased morbidity and mortality. BMC Cardiovasc Disord. 2019 Jun 10;19(1):139. doi: 10.1186/s12872-019-1117-0. PMID 31182031